CLINICAL TRIAL: NCT07283159
Title: Tenecteplase Plus Urinary Kallidinogenase for Acute Ischemic Stroke (TUKIS): a Prospective, Randomized, Double Blinded and Multi-center Study
Brief Title: Tenecteplase Plus Urinary Kallidinogenase for Acute Ischemic Stroke (TUKIS)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: General Hospital of Shenyang Military Region (Other)
Responsible Party: Principal Investigator, Hui-Sheng Chen, Director, General Hospital of Shenyang Military Region
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Y (2025) 357
Record Dates: First submitted 2025-12-02; First posted 2025-12-15 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Urinary Kallidinogenase with 0.15 PNA units dissolved in 100 ml of normal saline, administered via slow intravenous drip over no less than 50 minutes, once daily
  Interventions: Drug: Human Urinary Kallidinogenase
- Control group (Placebo Comparator): Urinary Kallidinogenase with placebo dissolved in 100 ml of normal saline, administered via slow intravenous drip over no less than 50 minutes, once daily
  Interventions: Drug: Human Urinary Kallidinogenase

INTERVENTIONS:
Drug: Human Urinary Kallidinogenase — Human Urinary Kallidinogenase is administered intravenously, with 0.15 PNA units dissolved in 100 ml of normal saline.

SUMMARY:
Human urinary kallidinogenase (HUK) is a tissue kallikrein extracted from human urine. Under certain conditions, tissue kallikrein can convert kininogen into kallidin and kinins, thereby promoting vascular endothelial function, and exerting anti-inflammatory and antioxidant effects. Preclinical and clinical studies have demonstrated that HUK can salvage the ischemic penumbra and significantly promote the establishment of collateral circulation. Existing research suggests that the combination of HUK with intravenous alteplase significantly improves neurological function in patients with acute ischemic stroke (AIS) without increasing the risk of hemorrhage. However, whether its combination with tenecteplase can further enhance neurological recovery in patients remains unreported. Based on the above discussion, this study aims to investigate the efficacy and safety of combining tenecteplase with HUK in the treatment of AIS.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 year;
* Acute ischemic stroke confirmed by neuroimaging;
* The time from last known well to treatment is within 4.5 hours;
* NIHSS ≥ 6 at randomization;
* Received intravenous tenecteplase (0.25mg/kg);
* First stroke onset or past stroke without obvious neurological deficit (mRS≤1);
* Signed informed consent.

Exclusion Criteria:

* Planed for endovascular treatment;
* Use of Edaravone Injection, Edaravone Dexborneol Injection, Butylphthalide Injection or Capsules after the onset of the current episode；
* Prior use of ACE inhibitors within a period less than 5 half-lives before the intended administration of Urinary Kallidinogenase for Injection；
* Pregnancy；
* Allergy to the investigational drug(s)；
* Comorbidity with other serious diseases;
* Participating in other clinical trials within 3 months;
* Patients not suitable for the study considered by researcher.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-01-20 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
proportion of excellent functional outcome (modified Rankin Scale (mRS) 0-1) | 90±7 days
  The minimum and maximum values of mRS are 0 and 6, respectively; higher score mean a worse outcome

SECONDARY OUTCOMES:
proportion of modified Rankin Scale (mRS) 0-2 | 90±7 days
  The minimum and maximum values of mRS are 0 and 6, respectively; higher score mean a worse outcome
ordinal distribution of modified Rankin Scale (mRS) | 90±7 days
  The minimum and maximum values of mRS are 0 and 6, respectively; higher score mean a worse outcome
change in National Institute of Health stroke scale (NIHSS) score | 24 (-6/+12) hours
  the minimum and maximum values of NIHSS are 0 and 42, respectively; higher NIHSS mean a worse outcome
change in National Institute of Health stroke scale (NIHSS) score | 10±2 days
  the minimum and maximum values of NIHSS are 0 and 42, respectively; higher NIHSS mean a worse outcome
occurrence of early neurological improvement (ENI) | 24 (-6/+12) hours
  ENI is defined as more than 4-point decrease in National Institute of Health stroke scale score
new stroke or other vascular event(s) | 90±7 days
symptomatic intracranial hemorrhage (sICH) | 24 (-6/+12) hours
  sICH was defined as any evidence of bleeding on the head computed tomographic scan associated with clinically significant neurological deterioration (≥4-point increase in NIHSS score).
major systemic bleeding events | 24 (-6/+12) hours
  Bleeding leading to a decrease in hemoglobin ≥ 2 g/dL or transfusion of ≥ 2 units of blood.
any bleeding events | 24 (-6/+12) hours
  Including skin and mucosal bleeding, gingival bleeding, bleeding at other organ sites, and other types of hemorrhage.
any intracranial hemorrhage | 10±2 days
  Heidelberg Bleeding Classification
all-cause mortality | 90±7 days
  death from any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurology, General Hospital of Northern Theater Command, Shenyang, China